CLINICAL TRIAL: NCT02004990
Title: Dental Office Prevention Strategies for Children: 10% Povidone Iodine (PI) Cleansing Prior to Fluoride Varnish (FV) Application
Brief Title: Dental Office Prevention Strategies for Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1310M44463; 8UL1TR000114-02 (NIH)
Record Dates: First submitted 2013-11-18; First posted 2013-12-09 (Estimated); Results first posted 2016-12-21 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Dental Plaque
Keywords: Children, Plaque
MeSH Terms: conditions — Dental Plaque; Plaque, Amyloid | interventions — Povidone-Iodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single cleansing procedure of 10% povidone iodine cleansing (Experimental): 10% povidone iodine cleansing
  Interventions: Procedure: Single cleansing procedure of 10% Povidone Iodine

INTERVENTIONS:
Procedure: Single cleansing procedure of 10% Povidone Iodine — Single cleansing procedure of 10% Povidone Iodine prior to an in-office 5% Sodium Fluoride varnish application

SUMMARY:
The overall goal of this study is to improve the standard of care in treating young children who often suffer from chronic caries (dental decay). Current standard of care for children under 12 years old includes a dental cleaning and fluoride treatment. Often this dental cleaning includes a 'dental prophylaxis' with a pumice based paste delivered by a small rubber-like cup that rotates on a slow-speed dental handpiece. The procedure of this dental prophylaxis removes the gross levels of plaque around the supragingival tooth surfaces. After this prophylaxis, a fluoride treatment is delivered. The National Maternal and Child Oral Health Resource Center at Georgetown University has published (Bertness J, Holt K) an extensive publication proving that 5% sodium fluoride varnish has become the 'standard of care' for fluoride treatment in children. This study includes this fluoride standard of care.

Prior to the administration of this standard of care fluoride treatment, a separate step of cleansing the tooth after the dental prophylaxis is added. This study uses a cleansing procedure of 10% povidone iodine (PI) cleansing prior to fluoride varnish (FV) application.

The primary aims of this study are:

1. to measure the changes in overall plaque levels after using a 10% povidone iodine (PI) cleansing prior to fluoride varnish (FV) application.
2. to measure the short term changes in the oral microbial ecology of dental plaque after 10% povidone iodine (PI) cleansing prior to fluoride varnish (FV) application.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria: Ages 6-12 years age. Recent history (< 24 months) of childhood caries, weight ≥ 15 kg, and current dental radiographic films within standard of care practices. At this time, we are looking for longitudinal changes within this cohort and are not using condition-matched controls.

Exclusion Criteria:

* Exclusion criteria: Weight <15 kg; Iodine or seafood allergy; hypersensitivity to fluoride varnish; antibiotics within the past 3 months; thyroid disease; significant past or current medical problem history, especially conditions that may affect salivary flow, dietary intake patterns, or routine oral hygiene.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jones, DDS, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Pediatric Dental Clinic, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Reilly C, Goettl M, Steinmetz M, Nikrad J, Jones RS. Short-term effects of povidone iodine and sodium fluoride therapy on plaque levels and microbiome diversity. Oral Dis. 2016 Mar;22(2):155-61. doi: 10.1111/odi.12407. Epub 2016 Jan 14. PMID 26662044

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Cleansing Procedure of 10% Povidone Iodine Cleansing
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Cleansing Procedure of 10% Povidone Iodine Cleansing
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Dental Plaque Levels Measures on Scale of 0-2
Description: Modified plaque index for the mixed dentition scale is 0-2 (0=best 2=worse)
Time Frame: 2-4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Cleansing Procedure of 10% Povidone Iodine Cleansing
Number analyzed (Participants) | 12
units on a scale | 0.391 (0.126)

2. Secondary Outcome: Dental Plaque Composition Measured by Numbers of Bacteria Present
Description: Dental plaque is a multispecies bacterial biofilm and the specific bacteria populating this biofilm will be measured. Measurement will be change in thickness of the biofilm
Time Frame: 2-4 weeks
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Single Cleansing Procedure of 10% Povidone Iodine Cleansing
Number analyzed (Participants) | 12
micrometers | 1.25 (.04)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Single Cleansing Procedure of 10% Povidone Iodine Cleansing
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes